CLINICAL TRIAL: NCT02358473
Title: Open-label, Multicenter Phase 1 Study of Mogamulizumab (KW-0761) in Combination With Docetaxel in Previously Treated Subjects With Non-small Cell Lung Cancer (NSCLC)
Brief Title: Study of Mogamulizumab + Docetaxel in Subjects With Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin, Inc. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0761-011
Record Dates: First submitted 2015-01-22; First posted 2015-02-09 (Estimated); Results first posted 2018-11-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Nonsmall Cell Lung Cancer; NSCLC; Non-Small-Cell Lung Carcinoma; Carcinoma, Non-Small Cell Lung; KW-0761; Mogamulizumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — mogamulizumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- mogamulizumab + docetaxel (Experimental): Mogamulizumab will be given as monotherapy in a 4-week run-in period. Subjects will then receive up to 6 cycles of mogamulizumab in combination with docetaxel at appropriate intervals.
  Subjects may then continue to receive mogamulizumab, at the same dose administered in Cycle 1, once every 3 weeks as monotherapy.
  Interventions: Biological: mogamulizumab; Drug: Docetaxel

INTERVENTIONS:
Biological: mogamulizumab — Mogamulizumab will be administered by IV infusion.
  Other Names: KW-0761; POTELIGEO®
Drug: Docetaxel — Docetaxel will be administered by IV infusion.
  Other Names: Taxotere; Docecad; DTX

SUMMARY:
The purpose of this study is to evaluate the safety of mogamulizumab in combination with docetaxel in adult subjects with previously treated locally advanced or metastatic non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed Stage IIIB or IV advanced or metastatic NSCLC with measurable neoplastic disease. Sputum cytology alone is not considered an acceptable method of diagnosis;
* Prior therapy must meet all of the following criteria:

  1. Subject has experienced disease progression or unacceptable toxicity/intolerance after receiving at least 1 systemic platinum-containing regimen;
  2. Subject with a tumor of non-squamous histology must be tested for epidermal growth factor receptor (EGFR) mutations and anaplastic lymphoma kinase (ALK) rearrangement. Subject with EGFR activating mutation or ALK rearrangement must have experienced disease progression or unacceptable toxicity/intolerance after receiving at least one EGFR tyrosine kinase inhibitor or ALK inhibitor;
  3. Subject has received PD-1/PD-L1 blockade or has been informed of the results of relevant positive Phase 3 trials with these agents.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1 at baseline;
* Minimum life expectancy of 3 months;
* Agrees to use a medically effective method of contraception. Male subjects and women of child-bearing potential (WOCBP) must agree to use effective contraception, e.g., oral contraceptives, double barrier method (condom plus spermicide or diaphragm plus spermicide), or practice true abstinence from sexual intercourse during the study and for 3 months after the last dose. Women of child-bearing potential include female subjects who have experienced menarche and have not undergone surgical sterilization or are not postmenopausal (defined as amenorrhea ≥ 12 consecutive months without an alternative medical cause);
* WOCBP must have a negative serum pregnancy test within 7 days prior to receiving investigational product and a negative urine pregnancy test on Day 1 of each Cycle;
* Recovered (i.e., Grade ≤ 1 or to a baseline level) from the effects of recent surgery, radiotherapy, chemotherapy, hormonal therapy, or other therapies for cancer (with the exception of alopecia for which no resolution is required and peripheral neuropathy which must have resolved to Grade ≤ 1 for subjects receiving prior taxane-based chemotherapy);
* Adequate organ function defined as below:

  1. Total bilirubin ≤ upper limit of normal (ULN);
  2. Hemoglobin (Hgb) ≥ 9.0 g/dL;
  3. Serum creatinine (sCr) ≤ 1.5 x ULN;
  4. Absolute neutrophil count (ANC) ≥ 1500 cells/mm3;
  5. Platelets ≥ 100 × 109/L;
* Sufficient archived tumor samples (if taken within 6 months prior to treatment may be submitted) available for PD assessments, or willingness to undergo a pre-treatment core needle biopsy, preferably of the primary tumor, in order to obtain such tissue;
* Willing and able to undergo a post-dose core needle biopsy.

Exclusion Criteria:

* Prior treatment with docetaxel or mogamulizumab;
* Requires administration of a prohibited medication or treatment;
* Has a significant uncontrolled intercurrent illness including, but not limited to:

  1. Ongoing or active infection requiring antibiotics;
  2. Clinically significant cardiac disease (class III, or IV of the New York Heart Association classification; unstable angina pectoris, myocardial infarction within 6 months or is post angioplasty or stenting within 6 months; clinically significant cardiac arrhythmia, or uncontrolled hypertension (i.e., systolic blood pressure > 150 mm Hg, diastolic blood pressure > 90 mmHg) despite anti-hypertensive medication;
  3. Uncontrolled diabetes, active liver disease, poorly controlled chronic obstructive pulmonary disease, serious or non-healing wound, ulcer, or fracture;
  4. Known or tests positive for human immunodeficiency virus, hepatitis B, or hepatitis C
  5. Active known auto-immune disease with the exception of autoimmune thyroiditis, vitiligo, and alopecia;
  6. Pleural effusion requiring repetitive drainage, i.e., an indwelling catheter or 2 thoracenteses with 6 weeks of the first dose of mogamulizumab;
* Received monoclonal antibodies (for any reason), chemotherapy, surgery, investigational therapy, or radiotherapy within 14 days of the first dose of mogamulizumab;
* Received live, attenuated vaccine within 28 days prior to the first dose of mogamulizumab;
* Use of immunosuppressive medication within 14 days before the first dose of mogamulizumab. Note: Inhaled, intranasal, intra-articular, or topical corticosteroids are allowed. Non-immunosuppresive doses of systemic steroids for adrenal replacement or for contrast allergy are allowed;;
* Any history or signs of central nervous system metastases;
* Any history or signs of pulmonary lymphangitic spread;
* Experienced a Grade 3 or higher hypersensitivity reaction to monoclonal antibodies or other therapeutic proteins, and the reaction could not be controlled or prevented on subsequent infusion with standard therapies such as antihistamines, 5-hydroxytryptamine (5-HT3) receptor antagonists, or corticosteroids;
* The subject has a history of severe hypersensitivity reactions to drugs formulated with polysorbate 80;
* History of second primary cancer within the past 5 years, with the exception of:

  1. Curatively resected non-melanomatous skin cancer;
  2. Curatively treated cervical intraepithelial neoplasia or prostate carcinoma with current prostate specific antigen (PSA) < 0.01 ng/mL; or
  3. Curatively treated ductal carcinoma in situ of the breast;
* The subject is pregnant or breastfeeding.
* The subject has aspartate aminotransferase and/or alanine aminotransferase > 1.5 × ULN, with concomitant alkaline phosphatase > 2.5 × ULN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kurman, Study Director — Kyowa Kirin, Inc.
Locations (5):
- United States (5):
  - Horizon Oncology, Lafayette, Indiana
  - John Hopkins University School of Medicine, Baltimore, Maryland
  - Gabrail Cancer Center Research, Canton, Ohio
  - MD Anderson, Houston, Texas
  - Cancer Therapy and Research Center, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Mogamulizumab + Docetaxel: Mogamulizumab (1.0 mg/kg, iv) was administered as monotherapy once weekly for 4 weeks. Subsequently, subjects received mogamulizumab (1.0 mg/kg) in combination with docetaxel (75 mg/m2), as separate infusions, on Day 1 every 3-weeks for up to 6 cycles.
Period: Overall Study
Arm/Group | Mogamulizumab + Docetaxel
Started | 13
Completed | 0
Not Completed | 13
Not completed — Disease Progession | 6
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Mogamulizumab + Docetaxel
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Adverse Events
Time Frame: Screening through 90 days after the last dose of study medication
Measure: Count of Participants; unit: Participants
Arm/Group | Mogamulizumab + Docetaxel
Number analyzed (Participants) | 13
Participants | 13

2. Primary Outcome: Number of Subjects Reporting Serious Adverse Events
Time Frame: Screening through 90 days after the last dose of study medication
Measure: Count of Participants; unit: Participants
Arm/Group | Mogamulizumab + Docetaxel
Number analyzed (Participants) | 13
Participants | 6

3. Primary Outcome: Number of Subjects Experiencing Dose-limiting Toxicity
Time Frame: First dose of study medications through 4 weeks after the last dose of study medication
Measure: Count of Participants; unit: Participants
Arm/Group | Mogamulizumab + Docetaxel
Number analyzed (Participants) | 13
Participants | 1

4. Secondary Outcome: Overall Response Rate
Description: The anti-tumor effect based on the Response Evaluation Criteria in Solid Tumors (RECIST version1.1), as well as by the immune-related RECIST (irRECIST).
Time Frame: One year
Population: A total of 6 subjects were excluded from the Efficacy Evaluable Set. Two (2) subjects did not have a baseline or post-baseline assessment for response; and 4 subjects were excluded due to "lack of investigational product(s) compliance", i.e., did not complete the first cycle of combination therapy (none of these subjects completed the Run-in period).
Measure: Count of Participants; unit: Participants
Arm/Group | Mogamulizumab + Docetaxel
Number analyzed (Participants) | 7
Participants | 0

5. Secondary Outcome: Progression Free Survival by RECIST 1.1
Description: as for outcome 4
Time Frame: One year
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Mogamulizumab + Docetaxel
Number analyzed (Participants) | 7
months | 1.87 [0.76 to 4.47]

6. Secondary Outcome: Overall Survival
Description: as for outcome 4
Time Frame: One year
Population: A total of 6 subjects were excluded from the Efficacy Evaluable Set. Two (2) subjects did not have a baseline or post-baseline assessment for response; and 4subjects were excluded due to "lack of investigational product(s) compliance", i.e., did not complete the first cycle of combination therapy (none of these subjects completed the Run-in period).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Mogamulizumab + Docetaxel
Number analyzed (Participants) | 7
months | 8.88 [2.70 to 8.88]

ADVERSE EVENTS:
Arm/Group | Mogamulizumab + Docetaxel
Serious Adverse Events (participants affected / at risk) | 6/13
Other Adverse Events (participants affected / at risk) | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mogamulizumab + Docetaxel (N=13)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2
Sepsis (Infections and infestations) | 2
Pneumonia Bacterial (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Hypotension (Vascular disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Renal failure actue (Renal and urinary disorders) | 1
Pyrexia (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mogamulizumab + Docetaxel (N=13)
Fatigue (General disorders) | 6
Nausea (Gastrointestinal disorders) | 5
Decreased appetite (Metabolism and nutrition disorders) | 4
Neutrophil count decreased (Blood and lymphatic system disorders) | 4
Pyrexia (General disorders) | 4
Diarrhea (Gastrointestinal disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Cardiac failure congestive (Cardiac disorders) | 2
Atrial fibrilliation (Cardiac disorders) | 2
Weight decreased (Metabolism and nutrition disorders) | 2
Orthostatic hypotension (Vascular disorders) | 2
Pneumonia (Infections and infestations) | 2
Sepsis (Infections and infestations) | 2
Neutropenia (Blood and lymphatic system disorders) | 2
Paraesthesia (Nervous system disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Pain (General disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Anxiety (Psychiatric disorders) | 1
Procedural site reaction (Injury, poisoning and procedural complications) | 1
Thrush (Infections and infestations) | 1
Mental status change (Psychiatric disorders) | 1
Hypertension (Vascular disorders) | 1
Palmer-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Insomnia (Psychiatric disorders) | 1
Asthenia (General disorders) | 1
Dizziness (Nervous system disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Deafness (Eye disorders) | 1
Balance disorder (Nervous system disorders) | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Chest pain (General disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Hypotension (Vascular disorders) | 1
Gout (Metabolism and nutrition disorders) | 1
Abdominal hernia (Gastrointestinal disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Platelet count decreased (Investigations) | 1
Post procedural oedema (Injury, poisoning and procedural complications) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Peripheral swelling (General disorders) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Oral candidiasis (Infections and infestations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Chills (General disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Disorientation (Psychiatric disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Local swelling (General disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Oedema peripheral (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No